CLINICAL TRIAL: NCT06464016
Title: Relapse of VAD Infections After Discontinuation of Anti-infective Therapies in Children.
Brief Title: Complications in Pediatric Mechanical Circulatory Assistance: Evaluation of Infection Management.
Acronym: VADINFECT
Status: Recruiting | Type: Observational
Sponsor: Claude Bernard University (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Lilot Marc, Official Director, Claude Bernard University
Other Study IDs: AGORA n°23-5221
Record Dates: First submitted 2023-10-10; First posted 2024-06-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Heart-Assist Devices; Infections; Heart Transplant Infection
MeSH Terms: conditions — Infections | interventions — Heart-Assist Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients with Berlin Heart EXCOR: Patient under 18 years old of age at the time of BH assistance in HCL Lyon France
  Interventions: Device: Ventricular Assist Device with Berlin Heart EXCOR

INTERVENTIONS:
Device: Ventricular Assist Device with Berlin Heart EXCOR — The Berlin Heart® EXCOR is a type of "artificial heart" pump that pulls blood from the ventricle and then sends that blood to the aorta or pulmonary trunc, thereby taking away extra work from the native heart. The device, which comes in several sizes, is not totally implanted inside the body.

SUMMARY:
Heart failure is a major cause of mortality and morbidity in children. Heart transplantation can significantly improve the prognosis of patients with severe heart failure, but access is limited by a shortage of transplants.

Long-term mechanical circulatory support is a major advance in the management of heart failure and can provide haemodynamic support while awaiting myocardial recovery or heart transplantation. The Berlin Heart (BH) EXCOR is the only long-term support system available for children.

Despite technical and medical advances in circulatory support, infection is a common complication and a major cause of morbidity and mortality in patients on BH.

There are few studies on the management of infection with mechanical support. Current ISHLT (International Society for Heart and Lung Transplantation) recommendations are based on expert opinion and observational studies. Some experts recommend anti-infective therapy until transplantation for specific support infections or for support-associated infections with persistent bacteraemia.

ELIGIBILITY:
Inclusion Criteria:

* patients under 18yo of age with Berlin Heart assisting device in Hospices Civils de Lyon, in France.

Exclusion Criteria:

* patients over 18 yo at the time of BH assistance
* unavailable documentation

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with terminal heart failure receiving BH assistance as bridge to transplant or bridge to recovery.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Relapse of VAD-infection after discontinuation of anti-infective therapy | 3 months
  Clinical and microbiological diagnosis of recurrence of infection with the same pathogen within 3 months of cessation of anti-infective therapy for a VAD-specific or VAD-related infection.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Panetta, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France